CLINICAL TRIAL: NCT03971357
Title: Prospective Randomized Study to Determine Whether Use of Rhopressa™ Accelerates Corneal Clearing After Removal of Descemet Membrane for Treatment of Fuchs Dystrophy
Brief Title: Trial of Netarsudil for Acceleration of Corneal Endothelial Restoration
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: variance of outcome measures was substantially greater than anticipated in the statistical plan
Sponsor: Price Vision Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-009
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2021-08

CONDITIONS: Fuchs' Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — netarsudil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Netarsudil (Experimental): Netarsudil ophthalmic solution 0.02%, dosed topically daily for the 3-month study duration or until 2 weeks after corneal clearing is complete, whichever occurs sooner
  Interventions: Drug: Netarsudil
- Placebo (Placebo Comparator): Placebo eye drop, dosed topically daily for the 3-month study duration or until 2 weeks after corneal clearing is complete, whichever occurs sooner.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Netarsudil — netarsudil opthalmic solution 0.02%
  Other Names: Rhopressa
  Arms: Netarsudil
Drug: Placebo — Placebo eye drops
  Arms: Placebo

SUMMARY:
Subjects with Fuchs dystrophy will be randomized to use either netarsudil or placebo eye drops to determine if the use of netarsudil accelerates migration of host peripheral corneal endothelial cells to restore the central endothelial cell layer.

DETAILED DESCRIPTION:
Subjects with Fuchs endothelial dystrophy will have the central corneal endothelium and guttae-covered Descemet membrane surgically removed. Subjects will be randomized to use netarsudil or placebo eye drops once daily. Visual acuity, corneal clearing and central endothelial cell density will be monitored for the 3-month study duration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient at least 18 years of age and of any race or ethnicity who is undergoing Descemet stripping only for Fuchs dystrophy
* Is able and willing to administer eye drops
* Is able to comprehend and has signed the Informed Consent form.

Exclusion Criteria:

* Active intraocular inflammation
* Corneal ulceration, keratitis, or conjunctivitis
* Known sensitivity to any of the ingredients in the study medications
* Abnormal eyelid function
* History of herpetic keratitis
* History of non-compliance with using prescribed medication
* Current or planned pregnancy within the study duration
* Concurrent involvement or participation in another randomized clinical trial within 30 days prior to enrollment in this study
* Any ocular or systemic condition (i.e., UNCONTROLLED systemic disease) or situation which in the investigator's opinion may put the patient at significant risk, confound the study results, or interfere significantly with the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, Jr, MD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arbelaez JG, Price MO, Price FW Jr. Long-term follow-up and complications of stripping descemet membrane without placement of graft in eyes with Fuchs endothelial dystrophy. Cornea. 2014 Dec;33(12):1295-9. doi: 10.1097/ICO.0000000000000270. PMID 25299425
- [Background] Moloney G, Petsoglou C, Ball M, Kerdraon Y, Hollhumer R, Spiteri N, Beheregaray S, Hampson J, D'Souza M, Devasahayam RN. Descemetorhexis Without Grafting for Fuchs Endothelial Dystrophy-Supplementation With Topical Ripasudil. Cornea. 2017 Jun;36(6):642-648. doi: 10.1097/ICO.0000000000001209. PMID 28476048
- [Background] Borkar DS, Veldman P, Colby KA. Treatment of Fuchs Endothelial Dystrophy by Descemet Stripping Without Endothelial Keratoplasty. Cornea. 2016 Oct;35(10):1267-73. doi: 10.1097/ICO.0000000000000915. PMID 27310885
- [Background] Soh YQ, Mehta JS. Regenerative Therapy for Fuchs Endothelial Corneal Dystrophy. Cornea. 2018 Apr;37(4):523-527. doi: 10.1097/ICO.0000000000001518. PMID 29384808
- [Background] Wacker K, Baratz KH, Bourne WM, Patel SV. Patient-Reported Visual Disability in Fuchs' Endothelial Corneal Dystrophy Measured by the Visual Function and Corneal Health Status Instrument. Ophthalmology. 2018 Dec;125(12):1854-1861. doi: 10.1016/j.ophtha.2018.06.018. Epub 2018 Aug 10. PMID 30104038

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Netarsudil | Placebo
Started | 10 | 9
Completed | 10 | 8
Not Completed | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Netarsudil | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10) | 58 (17) | 62 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Corneal Clearing After Endothelial Removal for Treatment of Fuchs Dystrophy
Description: The outcome measure was the percentage area of the cornea that remained edematous after removal of the endothelium. At the time of surgery, the surgeon recorded the lengths of the major and minor axes of the approximately circular area of endothelium removal; these values were used to calculate the area of stripping. At each postoperative exam, the examiner recorded the lengths of the major and minor axes of the edematous area; these values were used to calculate the area of edema. The percentage that remained edematous at 5 weeks was calculated by dividing the area of edema at 5 weeks by the area stripped.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: percentage of area stripped
Arm/Group | Netarsudil | Placebo
Number analyzed (Participants) | 10 | 9
percentage of area stripped | 42 (45) | 43 (49)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Netarsudil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 3/10 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Netarsudil (N=10) | Placebo (N=9)
cystoid macular edema (Eye disorders) | 1 (1) | 0 (0)
microcystic corneal epithelial bullae (Eye disorders) | 1 (1) | 0 (0)
eye discomfort (Eye disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT03971357/Prot_SAP_000.pdf